CLINICAL TRIAL: NCT02232152
Title: A Phase I Clinical Trial of Fluorouracil (5-FU) + CPI-613 Combination in Previously Treated Metastatic Colorectal Cancer Patients
Brief Title: CPI-613 and Fluorouracil in Treating Patients With Metastatic Colorectal Cancer That Cannot Be Removed by Surgery
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00028139; NCI-2014-01779 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CCCWFU #59314 (Other: Comprehensive Cancer Center of Wake Forest University); P30CA012197 (NIH)
Record Dates: First submitted 2014-09-02; First posted 2014-09-05 (Estimated); Last update posted 2023-08-07 (Actual); Status verified 2023-07

CONDITIONS: Mucinous Adenocarcinoma of the Colon; Mucinous Adenocarcinoma of the Rectum; Recurrent Colon Cancer; Recurrent Rectal Cancer; Signet Ring Adenocarcinoma of the Colon; Signet Ring Adenocarcinoma of the Rectum; Stage IIIA Colon Cancer; Stage IIIA Rectal Cancer; Stage IIIB Colon Cancer; Stage IIIB Rectal Cancer; Stage IIIC Colon Cancer; Stage IIIC Rectal Cancer; Stage IVA Colon Cancer; Stage IVA Rectal Cancer; Stage IVB Colon Cancer; Stage IVB Rectal Cancer
MeSH Terms: conditions — Colonic Neoplasms; Rectal Neoplasms | interventions — devimistat; Fluorouracil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (6,8-bis(benzylthio)octanoic acid, fluorouracil) (Experimental): Patients receive 6,8-bis(benzylthio)octanoic acid IV over 2 hours on days 1-4 and fluorouracil IV over 46 hours on days 2-4. Courses repeat every 2 weeks for 6 months in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: 6,8-bis(benzylthio)octanoic acid; Drug: fluorouracil; Other: pharmacological study; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: 6,8-bis(benzylthio)octanoic acid — Given IV
  Other Names: alpha-lipoic acid analogue CPI-613; CPI-613
Drug: fluorouracil — Given IV
  Other Names: 5-fluorouracil; 5-Fluracil; 5-FU
Other: pharmacological study — Correlative studies
  Other Names: pharmacological studies
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This pilot phase I trial studies the side effects and best dose of CPI-613 when given together with fluorouracil in treating patients with colorectal cancer that has spread to other parts of the body and cannot be removed by surgery. CPI-613 may kill tumor cells by turning off their mitochondria. Mitochondria are used by tumor cells to produce energy and are the building blocks needed to make more tumor cells. By shutting off these mitochondria, CPI-613 deprives the tumor cells of energy and other supplies that they need to survive and grow in the body. Drugs used in chemotherapy, such as fluorouracil, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Giving CPI-613 with fluorouracil may kill more tumor cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the maximum tolerated dose (MTD) of CPI-613 (6,8-bis[benzylthio]octanoic acid), when used in combination with 5-FU (fluorouracil), in patients with non-resectable metastatic colorectal cancer who have failed FOLFOX (leucovorin calcium, fluorouracil and oxaliplatin), FOLFIRI (leucovorin calcium, fluorouracil, and irinotecan hydrochloride) and, if Kirsten rat sarcoma viral oncogene homolog (KRAS) wild type, then a epidermal growth factor receptor (EGFR) inhibitor-based regimen.

SECONDARY OBJECTIVES:

I. To assess the pharmacokinetic (PK), safety and efficacy of various doses of CPI-613, when used in combination with 5-FU, in patients with non-resectable metastatic colorectal cancer.

OUTLINE: This is a dose-escalation study of 6,8-bis(benzylthio)octanoic acid.

Patients receive 6,8-bis(benzylthio)octanoic acid intravenously (IV) over 2 hours on days 1-4 and fluorouracil IV over 46 hours on days 2-4. Courses repeat every 2 weeks for 6 months in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 2 months for 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Histologically and cytologically confirmed metastatic colorectal adenocarcinoma (colon, rectal or colorectal cancer) that is not resectable
* Have failed or have not tolerated FOLFOX, FOLFIRI and, if KRAS wild type, then a EGFR inhibitor-based regimen
* Eastern Cooperative Oncology Group (ECOG) performance status being 0-2
* Women of child-bearing potential (i.e., women who are pre-menopausal or not surgically sterile) must use accepted contraceptive methods (abstinence, intrauterine device [IUD], oral contraceptive or double barrier device) during the study, and must have a negative serum or urine pregnancy test within 1 week prior to treatment initiation
* Fertile men must practice effective contraceptive methods during the study, unless documentation of infertility exists
* At least 2 weeks must have elapsed from any prior surgery
* Granulocyte count >= 1500/mm^3
* White blood cell (WBC) >= 3500 cells/mm^3 or >= 3.5 bil/L
* Platelet count >= 100,000 cells/mm^3 or >= 100 bil/L
* Absolute neutrophil count (ANC) >= 1500 cells/mm^3 or >= 1.5 bil/L
* Hemoglobin >= 9 g/dL or >= 90 g/L
* Aspartate aminotransferase (AST/serum glutamic oxaloacetic transaminase [SGOT]) =< 3 x upper normal limit (UNL), alanine aminotransferase (ALT/serum glutamate pyruvate transaminase [SGPT]) =< 3 x UNL (=< 5 x UNL if liver metastases present)
* Bilirubin =< 1.5 x UNL
* Serum creatinine =< 1.5 mg/dL or 13 umol/L
* International normalized ratio or INR must be =< 1.5 unless on therapeutic blood thinners
* No evidence of active infection and no serious infection within the past month
* Mentally competent, ability to understand and willingness to sign the informed consent form
* At least one measurable lesion as assessed by computed tomography (CT) scan using Response Evaluation Criteria in Solid Tumors (RECIST) criteria

Exclusion Criteria:

* Therapy with CPI-613 prior to participating in this trial
* Known hypersensitivity to 5-FU injection, poor nutritional state, known dipyrimidine dehydrogenase deficiency, or taking sorivudine (such as Usevir, brovavir, etc.)
* History of hypersensitivity to active or inactive excipients of any component of treatment
* Previous radiotherapy for central nervous system metastases
* Patients receiving any other standard or investigational treatment for their cancer, or any other investigational agent for any indication, within the past 2 weeks prior to initiation of treatment with study drugs
* Serious medical illness that would potentially increase patients' risk for toxicity
* Any active uncontrolled bleeding, and any patients with a bleeding diathesis (e.g., active peptic ulcer disease)
* History of abdominal fistula or gastrointestinal perforation =< 6 months prior to treatment with study drugs
* Pregnant women, or women of child-bearing potential not using reliable means of contraception
* Lactating females
* Fertile men unwilling to practice contraceptive methods during the study period
* Any condition or abnormality which may, in the opinion of the investigator, compromise the safety of patients
* Unwilling or unable to follow protocol requirements
* Symptomatic heart disease including but not limited to symptomatic congestive heart failure, symptomatic coronary artery disease, symptomatic angina pectoris, symptomatic myocardial infarction or symptomatic congestive heart failure
* Patients with a history of myocardial infarction that is < 3 months prior to registration
* Evidence of active infection, or serious infection within the past month
* Patients with known human immunodeficiency virus (HIV) infection, hepatitis B, or hepatitis C
* Patients who have received cancer immunotherapy of any type within the past 2 weeks prior to initiation of CPI-613 treatment; steroid use for management of refractory pain or for contrast induced allergy is allowed
* Requirement for immediate palliative treatment of any kind including surgery
* Any condition or abnormality which may, in the opinion of the investigator, compromise the safety of the patient

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2015-01-06 (Actual); Primary Completion 2019-02-19 (Actual); Study Completion 2023-01-11 (Actual)

PRIMARY OUTCOMES:
MTD of 6,8-bis(benzylthio)octanoic acid in combination with fluorouracil based on the incidence of dose-limiting toxicities graded according to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 4.0 | Up to 2 weeks

SECONDARY OUTCOMES:
Incidence of toxicity of 6,8-bis(benzylthio)octanoic acid and fluorouracil combination graded according to NCI CTCAE version 4.0 | Up to 3 years
  Examine toxicities by assessing each toxicity by grade.
PK parameters (maximum observed concentration, area under the curve, half-life, elimination rate constant, drug clearance, and volume of distribution) of 6,8-bis(benzylthio)octanoic acid in plasma samples | Week 1: days 1 and 4 before infusion of 6,8-bis(benzylthio)octanoic acid and at 30 minutes, 1, 1.5, 2, 4, 6 and 8 (optional) hours after the completion of infusion

OTHER OUTCOMES:
Progression-free survival (PFS) | Time from the first dose of 6,8-bis(benzylthio)octanoic acid to disease progression, assessed up to 3 years
  Plot a PFS curve using Kaplan-Meier methods, examine median PFS.
Overall response rate (ORR) (i.e., sum of complete response [CR] and partial response [PR]) | Up to 3 years
  Assess ORR and its 95% confidence interval.
Disease control rate (DCR) (i.e., sum of CR, PR, and stable disease) | Up to 3 years
  Assess DCR and its 95% confidence interval.

CONTACTS AND LOCATIONS:
Overall Officials: Caio Rocha Lima, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Comprehensive Cancer Center of Wake Forest University, Winston-Salem, North Carolina, United States

DOCUMENTS (1):
  • Informed Consent Form (2018-09-05): https://cdn.clinicaltrials.gov/large-docs/52/NCT02232152/ICF_000.pdf